CLINICAL TRIAL: NCT03273855
Title: Randomized Controlled Trial of Fecal Microbiota Transplantation in Severe Obesity
Acronym: RCTFMTOb
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University Hospital of North Norway (Other)
Collaborators: Norwegian University of Science and Technology (Other); Lovisenberg Diakonale Hospital (Other); Nordlandssykehuset HF (Other); Helse Nord (Industry); University of Tromso (Other); Norwegian University of Life Sciences (Other); University of Oslo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017/1655
Record Dates: First submitted 2017-08-31; First posted 2017-09-06 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Active Comparator. Transplant from Donor A or Donor B, or Donor C or Donore D, one transplant consist of 50-80g of feacal matter.
  Interventions: Other: Fecal microbiota transplantation
- Placebo (Placebo Comparator): Placebo. Patient will recieve an autologous fecal microbiota transplantation.
  Interventions: Other: Placebo: fecal microbiota transplantation

INTERVENTIONS:
Other: Fecal microbiota transplantation — The intervention treatment is fecal microbiota transplantation made of frozen donor feces. The FMT is transferred as rectal enema where we use a rectal probe with a balloon to prevent leakage and keep the solution long enough in the colon. The patient will stay on the bench in different positions for 20 minutes. We will encourage the participant to keep the solution in the colon as long as possible and give them four pills of loperamide before the procedure in order to reduce bowel motility.
  Arms: Intervention
Other: Placebo: fecal microbiota transplantation — The placebo group get fecal microbiota transplantation made of their own feces. The FMT is transferred as rectal enema where we use a rectal probe with a balloon to prevent leakage and keep the solution long enough in the colon. The patient will stay on the bench in different positions for 20 minutes. We will encourage the participant to keep the solution in the colon as long as possible and give them four pills of loperamide before the procedure in order to reduce bowel motility.
  Arms: Placebo

SUMMARY:
This is a randomized, double-blinded and placebo controlled prospective trial with sixty patients to investigate the effect of fecal microbiota transplantation (FMT) on body weight in patients with severe obesity. We will also collect data that possibly could give a better understanding of mechanisms of this correlation.

DETAILED DESCRIPTION:
Obesity is a main threat to public health in western countries. This condition increases the risk of developing type 2 diabetes, cardiovascular diseases, physical stress disorders, dispose for cancer and contributes to increased overall morbidity and mortality. However sustained weight loss lead to the reduction of risk factors and improvement of several obesity related co-morbidities.

Currently there are mainly two established treatments for severe obesity: a conservative approach through lifestyle intervention and a surgical approach with bariatric surgery. The gut microbiota is recognized as an environmental modulator of nutritional uptake and body weight. This has led to the hypothesis that the gut microbiota could be a therapeutic target fighting obesity. Fecal microbiota transplantation (FMT) has been applied for more than 50 years, and is a established treatment for refractory recurrent infection with Clostridium Difficile (CDI). Recent scientific studies have also applied FMT as treatment for other diseases like inflammatory bowel disease, irritable bowel disease and even metabolic syndrome and the results are promising.

The sample size is determined based on data from the outpatient clinic at UNN Harstad medical department. Patients here have an average weight loss of 2,5 % with conservative treatment. This will therefore be the expected result in the control group (receiving placebo). A weight reduction of 5-10% leads to significant improvement of health and quality of life, and a weight change of this magnitude is therefore the hypothesis. The difference between the two groups is estimated to 7,5 %. With these historical results, the sample size is estimated to be 19 patients in each group. Extreme values will be eliminated; more than 3 SD out of the average in the group. In this patient group, we must also be prepared to high degree loss of follow-up near one third, which is also the experience from the clinic. We will include totally 60 patients, 30 in each group.

The investigators are planning a randomized, double-blinded and placebo controlled prospective trial with sixty patients to investigate the effect of fecal microbiota transplantation (FMT) on body weight in patients with severe obesity. In the trial there will also be collected data that possibly could give a better understanding of mechanisms of this correlation; with insulin resistance, blood pressure, complete body scan, inflammation and biochemical parameters of hepatic steatosis, changes in the patients microbiota and the development in quality of life as secondary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 40 or BMI > 35 kg/m2 combined with comorbidity related to obesity.

Exclusion Criteria:

* Symptomatic cardiovascular disease, lung disease, cirrhosis or significant renal failure.
* Patients who are pregnant or breastfeeding
* Patients who have a confirmed malignancy or cancer
* Patients who are immunocompromised
* Previous gastric or small intestinal surgery that alters gut anatomy such as fundoplication, gastric resection, gastric bypass, small bowel resection, and ileoectomy
* Established drug- or alcohol abuse or particularly unstable psychosocial circumstances.
* History of cholecystektomy (gut microbiota composition could be affected by bile acid composition)
* New drugs the last three months or during the follow-up period that can impact on metabolism or body weight
* Antibiotic treatment the last three months

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-05-13 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in individual weight loss (kg). | Change from baseline body weight at 12 months post FMT
  Partisipants will be measured at the outpatient clinic, medical department UNN Harstad, and weight in kilograms (kg) will be recorded. The data will be represented both as average weight change and as bar charts with >10%, with comparison between the intervention and control group.
  Chi Square or Fischer exact test will be used to present responders and non-responders in the active and controll group. We will use odds ratio to present responders in the active group.

SECONDARY OUTCOMES:
Change in individual weight loss (kg) | Change from baseline body weight at 3, 6 and 12 months after FMT
  Partisipants will be measured at the outpatient clinic, medical department UNN Harstad, and weight in kilograms (kg) will be recorded. The data will be represented both as average weight change and as bar charts with >5%, >15% and >20% weight loss, with comparison between the intervention and control group at each controll point.
  Chi Square or Fischer exact test will be used to present responders and non-responders in the active and controll group. We will use odds ratio to present responders in the active group.
Change in waist circumference (cm) | Change from baseline waist circumferense at 3, 6 and 12 months after FMT
  Participants will be measured at the outpatient clinic, medical department UNN Harstad, and waist circumference (cm) will be recorded.
Changes in HbA1c (mmol/mol) | Change from baseline HbA1c at 3, 6 and 12 months after FMT
  Together with C-peptide, fasting glucose and insuline it will be used to research insuline resistance.
Changes in fasting glucose (mmol/L) | Change from baseline fasting glucose at 3, 6 and 12 months after FMT
  Together with HbA1c, C-peptide, and insuline it will be used to research insuline resistance and calculate HOMA-IR and HOMA-B
Changes in insuline (pmol/L) | Change from baseline insuline at 3, 6 and 12 months after FMT
  Together with HbA1c, C-peptide, and fasting glucose it will be used to research insuline resistance and calculate HOMA-IR and HOMA-B
Changes in C-peptide (pmol/L) | Change from baseline C-peptide at 3, 6 and 12 months after FMT
  Together with HbA1c, fasting glucose and insuline it will be used to research insuline resistance.
Change in blood pressure | Change from baseline blood pressure at 3, 6 and 12 months after FMT
  Participants blood pressure (mmHg) will be measured at the outpatient clinic, medical department UNN Harstad. Blood pressure is collected as the average of the last two out of three measurements, at the end of 5 min resting period in supine position.
Change in sedimentation rate (mm/t) | Change from baseline sedimentation rate at 3, 6 and 12 months after FMT
  We will measure sedimentation rate, and together with hs-CRP and cytokine panel we will investigate inflamation between the group recieving placebo and the group recieving active transplant.
Change in hs-CRP (mg/L) | Change from baseline hs-CRP at 3, 6 and 12 months after FMT
  We will measure hs-CRP, and together with sedimentation rate and cytokine panel we will investigate inflamation between the group recieving placebo and the group recieving active transplant.
Changes in multiplex cytokine panel (pg/mL) | Change from baseline cytokine panel at 3, 6 and 12 months after FMT
  We will run a multiplex cytokinepanel consiting of 27 different cytokines to see if the consentration of blood cytokines changes in participants after active treatment/placebo. The cytokine panel consists of TNF-a, IFN-g, IL-1b, IL-1ra, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-9, IL-10, IL-12(p70), IL-13, IL-15, IL-17A, MCP-1(MCAF), IP-10, Eotaxin, MIP-1a, MIP-1b, RANTES, G-CSF, GM-CSF, Basic FGF, PDGF-BB, VEGF.
Changes in biochemical parameters of hepatic steatosis (U/L) | Change from baseline biochemical parameters at 3, 6 and 12 months after FMT
  Photometric analysis. We will measue AST, ALT, ALP, ɣGT and amylase to look at changes in biochemical parameters of hepatic steatosis between the group recieving placebo and the group recieving active transplant
Changes in lipid profile based on HDL/LDL (mmol/L) and cholesterol (mmol/L) | Change from baseline lipid profile at 3, 6 and 12 months afterFMT
  Photometric analysis. Changes in cholesterol and HDL/LDL be used to look at changes in lipid profile between the group recieving placebo and the group recieving active transplant
Changes in life quality measured using RAND-36 questionnaire | Change from baseline RAND-36 score 12 months after FMT
  RAND-36- Item Short Form Health Survey. The SF-36 consists of eight scaled scores (vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health), which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. By an independent sample T-test (or, if necessary, non-parametric Mann-Whitney) we will compare change in global score. We will apply last value forward for missing values
Changes in psychiatric comorbidity measured by HSCL-25 | Change from baseline HSCL-25 score 12 months after FMT
  HSCL-25. Consists of 25 questions. Each answer to a question has a value of 1-4. A total score over 1,75 points to psychological issues or impaired mental health
Changes in dietary intake measured by FFQ | Change from baseline FFQ score at 3, 6 and 12 months after FMT
  FFQ Change in dietary intakes measured using Food Frequency Questionnaire at baseline and at 3, 6 and 12 months after FMT will be examined.
  Energy measured as kcal, nutrition (gram) and different food groups reported as gram/day
Changes in life style measured by IPAQ | Change from baseline IPAQ score at 3, 6 and 12 months after FMT
  IPAQ Categorical Score
  Three levels (categories) of physical activity are proposed:
  Category 1: Low This is the lowest level of physical activity. Those individuals who not meet criteria for categories 2 or 3 are considered low/inactive.
  Category 2: Moderate
  Any one of the following 3 criteria:
  * 3 or more days of vigorous activity of at least 20 minutes per day OR
  * 5 or more days of moderate-intensity activity or walking of at least 30 minutes per day OR
  * 5 or more days of any combination of walking, moderate-intensity or vigorous intensity activities achieving a minimum of at least 600 MET-min/week.
  Category 3: High
  Any one of the following 2 criteria:
  * Vigorous-intensity activity on at least 3 days and accumulating at least 1500 MET-minutes/ week OR
  * 7 or more days of any combination of walking, moderate-intensity or vigorous intensity activities achieving a minimum of at least 3000 MET-minutes/week
Gut microbiota composition and function | Change from baseline microbiota composition at 3, 6 and 12 months after FMT
  Microbiota analysis and SCFA in faeces
Short difficult childhood questionnaire | At baseling
  Questions of childhood trauma, four or six questions
Childhood trauma Questionnaire (CTQ) | Once during the follow up period in the study
  A validated questionnaire to collect self-reported data about adverse childhood experiences
Heart rate variability (HRV) | HRV will be measured at inclusion and 3.months post FMT
  A dysbiotic gut microbiota that signals with the vagal nerve can cause an exaggerated stress response in obesity characterised by decrease in heart rate variability.

OTHER OUTCOMES:
Engraftment of donor microbiota at 1, 3, 6 and 12 months. | Inclusion, 2, 3, 6 and 12 months after FMT
  Comparison between baseline profile, post FMT and donor profile will show if engraftment of donor microbiota parallels clinical response to active FMT.
Eating behaviour | Change from baseline binge eating questionnaore score 12 months after FMT
  Binge eating questionnaire
Questionnaire about the impact of covid-19 on life style changes and eating habits | Once during the follow up period in the study
  Participants which had undergone intervention and were in the follow up period, had all their appointments at the obesity clinic at UNN Harstad canceled, due to the covid-19 outbreak in the period march-20 to juli-20. This might have impacted their weight loss motivation and life style changes. We therefore asked them five questions, which we hope will shed light on the challenges they might encountered during the period of restrictions implemented by the Norwegian government.

CONTACTS AND LOCATIONS:
Overall Officials: Per C Valle, PhD, Principal Investigator — University Hospital of North of Norway; Maria S Fjellstad, cand.med, Study Chair — University Hospital of North of Norway; Hege M Hanssen, M.Sc, Study Chair — University Hospital of North Norway
Locations (1):
- University Hospital of North Norway, Harstad, Troms, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hanssen HM, Fjellstad MS, Skjevling L, Johnsen PH, Kulseng B, Goll R, Alma KH, Valle PC. Randomised, placebo-controlled, double-blinded trial of fecal microbiota transplantation in severe obesity: a study protocol. BMJ Open. 2023 Dec 27;13(12):e073242. doi: 10.1136/bmjopen-2023-073242. PMID 38151280